CLINICAL TRIAL: NCT01628458
Title: Phase II Study: Radiofrequency Ablation of Locally Advanced Pancreatic Cancer
Brief Title: Safety Study of Radiofrequency Ablation of Locally Advanced Pancreatic Cancer
Acronym: RFA of LAPC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, R. van Hillegersberg, Professor in surgery, UMC Utrecht
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-018
Record Dates: First submitted 2012-06-20; First posted 2012-06-26 (Estimated); Last update posted 2015-02-02 (Estimated); Status verified 2015-01

CONDITIONS: Locally Advanced Pancreatic Cancer
Keywords: Pancreatic cancer; locally advanced; irresectable; Radiofrequency; RFA
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- radiofrequency ablation (Experimental)
  Interventions: Procedure: radiofrequency ablation (RFA)

INTERVENTIONS:
Procedure: radiofrequency ablation (RFA) — RFA with CELON bipolar probes. Settings: Power 30 watts, total energy 15 KJ.
  Other Names: CELON Power System, CE mark 0197

SUMMARY:
The purpose of the study is to determine the safety of radiofrequency ablation of locally advanced pancreatic cancer that can not be surgically removed with the current standard procedures. Complications after the operation will be registered. Moreover a pain score will be determined, length of hospital stay, chemotherapy, survival, progression free survival and a tumour marker.

DETAILED DESCRIPTION:
Pancreatic cancer is the fourth leading cause of cancer related death in the Western world. At time of diagnosis, 20% of patients present with a resectable tumour, 40% with an irresectable locally advanced tumour (without metastases) and 40% with metastatic disease. The median survival of patients with irresectable locally advanced pancreatic cancer is only 6 months. Currently, there is no effective treatment for these patients. Therefore, there is an urgent need for new therapies. Radiofrequency ablation (RFA) is a technique that has been demonstrated to be effective in the treatment of several irresectable tumours. RFA produces local tumour destruction through high frequency alternating current flowing from an electrode implanted directly into the tumour and causing frictional heating. The purpose of this study is to determine the safety of RFA-pancreas in patients with non-metastasized, irresectable, locally advanced pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with irresectable locally advanced pancreatic cancer found at laparotomy with histologic diagnosis before start of RFA
2. Patient considered eligible to undergo pancreatic surgery as assessed by the general criteria of the departments of anaesthesiology and surgery of the UMC Utrecht
3. Fully informed written consent given

Exclusion Criteria:

1. Patients younger than 18 years
2. Pregnancy
3. Patients with distant metastases
4. Portal vein thrombosis seen on CT preoperatively

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2012-09; Primary Completion 2014-07 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Safety | Within 30 days after the RFA procedure
  The safety will be specified as the percentage of patients with complications directly related to RFA and the routinely performed double-bypass procedure, requiring re-intervention (i.e. endoscopy, radiology, or surgery). This is also known as a complication of grade III or higher in the Clavien-Dindo classification (internationally accepted classification for surgical complications). Moreover all in-hospital complications or complications developed within 30 days after the RFA procedure will be evaluated according to the Clavien-Dindo classification.

SECONDARY OUTCOMES:
survival | 2 years after RFA procedure
VAS pain score | 3 months
length hospital stay | 3 months
progression free survival | 2 years after RFA procedure
CA19-9 response | 2 years after RFA procedure
Chemotherapy | 2 years
  Type, frequency, dosage and duration of chemotherapy will be registered.

CONTACTS AND LOCATIONS:
Overall Officials: Richard van Hillegersberg, Professor, Principal Investigator — UMC Utrecht
Locations (1):
- University Medical Center Utrecht, Utrecht, Utrecht, Netherlands

REFERENCES:
- [Background] Cantore M, Girelli R, Mambrini A, Frigerio I, Boz G, Salvia R, Giardino A, Orlandi M, Auriemma A, Bassi C. Combined modality treatment for patients with locally advanced pancreatic adenocarcinoma. Br J Surg. 2012 Aug;99(8):1083-8. doi: 10.1002/bjs.8789. Epub 2012 May 30. PMID 22648697
- [Background] Girelli R, Frigerio I, Salvia R, Barbi E, Tinazzi Martini P, Bassi C. Feasibility and safety of radiofrequency ablation for locally advanced pancreatic cancer. Br J Surg. 2010 Feb;97(2):220-5. doi: 10.1002/bjs.6800. PMID 20069610